CLINICAL TRIAL: NCT03355456
Title: Prospective, Multi-center, Randomized, Evaluation Comparing the Protocol Specified Ablation Approach to the Current Standardized Ablation Approach in the Treatment of Non-paroxysmal Atrial Fibrillation.
Brief Title: Low Voltage-Directed Catheter Ablation for Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohad Ziv (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ohad Ziv, Director, Cardiac Electrophysiology, Principal Investigator, Professor of Medicine, MetroHealth Medical Center
Organization: MetroHealth Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB17-00025
Record Dates: First submitted 2017-11-16; First posted 2017-11-28 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation - Symptomatic
Keywords: Persistent atrial fibrillation; Medication refractory atrial fibrillation; Pulmonary vein isolation procedure; Low voltage directed ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomized comparison of two ablation techniques:
  1. Pulmonary vein isolation (PVI) alone to
  2. PVI plus total left atrial low voltage-directed ablation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to whichever ablation arm they are randomized to. Events adjudicator will be blinded to randomization arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation (PVI) alone (Active Comparator): Radiofrequency ablation procedure to isolate pulmonary veins without other intervention performed..
  Interventions: Procedure: Radiofrequency ablation
- PVI+Total LT Atrial low voltage ablation (Active Comparator): PVI radiofrequency ablation along with ablation of areas of "low voltage" identified.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Ablation procedure to eliminate atrial fibrillation
  Other Names: Pulmonary vein isolation, low-voltage ablation

SUMMARY:
A two-pronged approach to evaluate long term success of non-paroxysmal ablation when using a:

1. specified low voltage-directed with pulmonary vein isolation (LD+PVI) approach compared to ,
2. an approach of pulmonary vein isolation (PVI) alone.

DETAILED DESCRIPTION:
Patients that meet both inclusion and exclusion criteria will be randomized by the study clinical center upon determination of low-voltage being present using 3-D mapping during index. Enrolled subjects who do not have low voltage will be followed in a registry and their data will be evaluated separately. Low-voltage patients will be randomized 1:1 into one of the following arms:

* PVI with additional total left atrial low voltage-directed ablation.
* PVI alone.

All patients will receive the best conventional medical therapy and anticoagulation use based upon HRS consensus recommendations taking into account their baseline risk factors for stroke. The need for interruption of anticoagulation and antiarrhythmic drug therapy for the procedure will be determined by the operator and their center guidelines.

The trial requires continuous monitoring for atrial arrhythmias. Investigators will recommend the use of implantable loop recorders (ILR) but continuous 30 day monitoring with auto-trigger function may be substituted at the 6, 9 and 12 month time points. The ILR device will be implanted under sterile conditions at the manufacture's recommended site on the precordium for arrhythmia monitoring. Implantation will occur between 1 month prior and 3 months post ablation since there will be a 3 month post ablation blanking period. If a dual chamber device is already present, implantation will not be required. iWatch, Kardia or other non-FDA approved cardiac monitoring can be used to preliminarily identify AF recurrence but AF recurrence must be separately verifiable by ECG or other FDA-certified monitoring system.

One year follow-up is planned. Post procedure care is per standard of care with follow-up at 1 month, 3 months, 6 months, 9 months and 12 months. ECG at every follow-up is performed. Download of arrhythmia data will occur at each of these visits as well. Investigators will use the typical post ablation blanking period for recurrence of atrial fibrillation of 3 months. Antiarrhythmic medications can be used during the typical "blanking period" of 3 months post procedure. But per protocol are stopped at 3 months post procedure (2 months post procedure in case of amiodarone).

Investigators will compare time freedom from first arrhythmia event, defined as a sustained episode of atrial fibrillation or atrial tachycardia. Secondary endpoints will be compared as well (see secondary end point defined). Re-initiation of an antiarrhythmic drug after 3 months will be considered a failure of primary endpoint of arrhythmia free survival. However, Anti-arrhythmic medication use after the blanking period for ventricular arrhythmias will not be included as an event. Anticoagulation is continued and monitored based on previous guidelines with use stratified by baseline stroke risk. A recording (CD) of the mapping during the procedure is to be obtained and retained for possible future analysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Non-Paroxysmal Atrial Fibrillation.
2. Failed or intolerable to at least 1 one antiarrhythmic drug (AAD).
3. 18-85 year of age at time of consent.
4. Scheduled to undergo a clinically indicated AF ablation procedure.
5. Able and willing to comply with all protocol visit requirements.
6. Signed Patient Informed Consent (ICF).
7. Presence of low voltage in the left atrium on 3-D map during index catheter ablation procedure

Exclusion Criteria:

Subjects will be excluded if any of the follow criteria are present:

1. History of prior left-sided catheter or surgical ablation for AF or atypical atrial flutter, including MAZE or mini MAZE.

   * Prior ablation for typical atrial flutter or left-sided ablation for WPW, AV node reentry tachycardia or focal ectopic atrial tachycardia may be included.
2. Uncontrolled heart Failure or NYHA Class IIIb or IV heart failure.
3. Ejection Fraction < 0.20.
4. Active ventricular tachycardia requiring treatment with catheter ablation or anti-arrhythmic drug within the last 6 months.
5. Left atrial size > 60 mm diameter on echocardiogram.
6. "Long standing" persistent AF defined as > or = 1 year of continuous atrial fibrillation at the time of enrollment.
7. Severe pulmonary hypertension (PAP > 70 mmHg)
8. Unstable valvular disease.
9. AF secondary to electrolyte imbalance, thyroid disease or reversible non- cardiac cause.
10. Poor candidate for general anesthesia.
11. Anticipated survival < 1 year.
12. MI or CABG within 3 months.
13. Left atrial thrombus in pre-procedure imaging within 4 weeks of the ablation procedure.
14. Any documented thromboembolic event within 6 months of the ablation procedure.
15. Contraindication to anticoagulation.
16. Inability to have implantable monitoring device for atrial fibrillation burden with no pre-existing cardiac device that can monitor atrial arrhythmias OR inability to wear external Holter Monitor continuously for 4 weeks.
17. Significant congenital anomaly or medical condition that may affect the integrity of study data.
18. Women who are pregnant - pregnancy test required if pre-menopausal or non-sterile.
19. Active enrollment in another investigational study involving a drug or device.
20. Inability to undergo complete voltage mapping in normal sinus rhythm - see intraprocedural protocol.
21. Presence of any medical or psychological condition or medical non-compliance history that may adversely impact study outcomes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-07-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from first arrhythmia recurrence defined as sustained symptomatic or asymptomatic atrial fibrillation, atrial flutter or atrial tachycardia. | Any event between the 3 month blanking period and 1 year post-ablation.
  The primary endpoint is freedom from sustained symptomatic or asymptomatic atrial arrhythmia (atrial fibrillation, atrial flutter or atrial tachycardia - AT/AF) i.e.; NO change from sinus rhythm to atrial arrhythmia between 3 -12 months after ablation. Recurrence of AF/AT excludes the 3 month blanking period. Sustained AF/AT is defined as >30 seconds as recorded on a monitoring device.

SECONDARY OUTCOMES:
Reduced arrhythmia burden (frequency that arrhythmia occurs). | Between the 3 month blocking period and 1 year post-ablation.
  Comparison of arrhythmia burden as determined by the composite percent of atrial arrhythmia during the total time recorded on implantable monitoring devices.
Freedom from sustained AF/AT | Any event between the 3 month blocking period and 1 year post-ablation.
  Freedom from sustained AF/AT is defined as >30 seconds as recorded on a monitoring device.
Freedom from any symptomatic AF/AT | Any event between the 3 month blocking period and 1 year post-ablation.
  Freedom from any symptomatic AF/AT is defined regardless of duration as recorded on a monitoring device.
Reduced need for antiarrhythmic drugs (AAD) | Any event between the 3 month blocking period and 1 year post-ablation.
  Comparison of the use of AAD therapy to control atrial arrhythmias after a successful ablation.

OTHER OUTCOMES:
Incidence of procedure related adverse events. | Any event up to 1 year post-ablation.
  The safety endpoint is the incident of procedure related adverse events comparing the 3 arms of the study. Adverse events being tracked are:
  1. All-cause mortality
  2. Atrio-esophageal fistula (through 12 mo)
  3. Atrial perforation
  4. Cardiac Tamponade
  5. Pericardial Effusion
  6. Pericarditis
  7. Heart Block
  8. Myocardial infarction
  9. Cerebrovascular Accident (CVA)
  10. Transient ischemic Attack
  11. Thromboembolism
  12. PV stenosis >70% from baseline (through 12 mo)
  13. Diaphragm Paralysis
  14. Pulmonary Edema
  15. Pneumothorax
  16. Limb Paralysis
  17. Procedural blood loss ≥ 1000cc
  18. Respiratory failure
Tertiary endpoints | Any event up to 1 year post-ablation.
  For patients not randomized, data will be collected for the same endpoints as randomized patients. Additionally, data on atrial ERP and location of additional ablation that will be collected will be used in arrhythmia recurrence analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Ziv, MD, Principal Investigator — MetroHealth System, Ohio
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. J Interv Card Electrophysiol. 2012 Mar;33(2):171-257. doi: 10.1007/s10840-012-9672-7. PMID 22382715
- [Background] Themistoclakis S, Raviele A, China P, Pappone C, De Ponti R, Revishvili A, Aliot E, Kuck KH, Hoff PI, Shah D, Almendral J, Manolis AS, Chierchia GB, Oto A, Vatasescu RG, Sinkovec M, Cappato R; Atrial Fibrillation Survey Investigators. Prospective European survey on atrial fibrillation ablation: clinical characteristics of patients and ablation strategies used in different countries. J Cardiovasc Electrophysiol. 2014 Oct;25(10):1074-81. doi: 10.1111/jce.12462. Epub 2014 Jul 8. PMID 24891043
- [Background] Lin YJ, Chang SL, Lo LW, Hu YF, Chong E, Chao TF, Chung FP, Liao J, Li CH, Tsao HM, Kao T, Chen YY, Huang JL, Chen SA. A prospective and randomized comparison of limited versus extensive atrial substrate modification after circumferential pulmonary vein isolation in nonparoxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2014 Aug;25(8):803-812. doi: 10.1111/jce.12407. Epub 2014 Apr 9. PMID 24628987
- [Background] Nademanee K, McKenzie J, Kosar E, Schwab M, Sunsaneewitayakul B, Vasavakul T, Khunnawat C, Ngarmukos T. A new approach for catheter ablation of atrial fibrillation: mapping of the electrophysiologic substrate. J Am Coll Cardiol. 2004 Jun 2;43(11):2044-53. doi: 10.1016/j.jacc.2003.12.054. PMID 15172410
- [Background] Hwang C, Chen PS. Ligament of Marshall: why it is important for atrial fibrillation ablation. Heart Rhythm. 2009 Dec;6(12 Suppl):S35-40. doi: 10.1016/j.hrthm.2009.08.034. PMID 19959141

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT03355456/Prot_SAP_000.pdf